CLINICAL TRIAL: NCT05416372
Title: Engaging Religious Leaders to Reduce Blood Pressures in Tanzanian Communities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-06023670; R01HL161673 (NIH)
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: Religious Leaders; Community Engagement; Hypertension; Tanzania
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: 20 communities will be stratified by population size (< or ≥ 20,000) and randomly ordered within strata using a computerized random number generator. A statistician will generate a list of all of possible random permutations that allocate equal numbers of communities from each stratum to the intervention and to the control. Investigators will then invite two representatives from each of the 20 communities to a public randomization ceremony. During this ceremony, representatives will blindly choose numbered tennis balls from an opaque bag to identify the permutation of allocations that will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control communities (No Intervention): Communities randomized to the control arm will receive a strengthening of the capacity to manage blood pressure at their local health center. Healthcare workers at the local health center will receive standard supplies, reference materials, and training in blood pressure measurement and management on-site. In the event of any stock-outs due to higher demand for antihypertensives during the trial implementation, the trial will temporarily provide these medications to primary health facilities until the Ministry of Health supply chain is restored. Of note, control communities will receive Religious Engagement in Health Intervention after the trial is complete.
- Religious Engagement in Health Intervention communities (Experimental): Communities randomized to the intervention arm will receive a strengthening of the capacity to manage blood pressure at their local health center plus Religious Engagement in Health Intervention for blood pressure (BP), which includes three evidence-based components; 1) educational sessions for Christian and Muslim leaders on religious teachings and medical aspects of BP, 2) equipping religious leaders to provide BP teaching in their communities using knowledge learned from educational sessions and through longitudinal mentorship meetings, and 3) community BP screening organized by religious leaders in partnership with local health care workers, and referrals for clinical care as needed.
  Interventions: Behavioral: Religious Engagement in Health Intervention

INTERVENTIONS:
Behavioral: Religious Engagement in Health Intervention — Religious Engagement in Health Intervention for blood pressure (BP) includes three evidence-based components: (1) educational sessions for Christian and Muslim leaders on religious teachings and medical aspects of BP, (2) equipping religious leaders to provide BP teaching in their communities using knowledge learned from educational sessions and through longitudinal mentorship meetings, and (3) community BP screening organized by religious leaders in partnership with local health care workers, and referrals for clinical care as needed.
  Arms: Religious Engagement in Health Intervention communities

SUMMARY:
The investigators hypothesize that communities in which religious leaders are provided with education about blood pressure and how to measure blood pressure will have lower overall average blood pressures than communities in which religious leaders do not receive education about blood pressure.

DETAILED DESCRIPTION:
This research is being done to determine whether the Religious Engagement in Health Intervention can reduce community blood pressure. The study is being conducted in the Northwestern Tanzania. 20 communities will be involved: 10 will be randomized to the Religious Engagement in Health Intervention arm, and 10 will be randomized to the control arm. The Religious Engagement in Health Intervention includes the following three evidence-based components: (1) educational sessions for Christian and Muslim leaders on religious teachings and medical aspects of blood pressure, (2) equipping religious leaders to provide blood pressure teaching in their communities using knowledge learned from educational sessions and through longitudinal mentorship meetings, and (3) community blood pressure screening organized by religious leaders in partnership with local health care workers, and referrals for clinical care as needed.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥35 years of age
* Has lived in the community for ≥1 year
* Household identified for random sampling is primary residence: has slept in the household at least once in the past 2 weeks and considers this their primary residence

Exclusion Criteria:

* First-degree relative from the same household already enrolled
* Relative of the same sex from the same household already enrolled

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24000 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in community systolic blood pressure | Baseline; 12months
  Before and 12 months after the intervention, investigators will estimate the true mean community BP by sampling 400 randomly selected adult community members (age ≥35 years) in each of the 20 communities.

SECONDARY OUTCOMES:
Change in awareness of hypertension | Baseline; 12 months
  Change in the percent of people with hypertension who are aware that they have hypertension, from baseline to 12 months
Change in awareness of hypertension | Baseline; 24 months
  Change in the percent of people with hypertension who are aware that they have hypertension, from baseline to 24 months
Change in treatment of hypertension | Baseline; 12 months
  Change in percent of people with hypertension who are on treatment for hypertension, from baseline to 12 months
Change in treatment of hypertension | Baseline; 24 months
  Change in percent of people with hypertension who are on treatment for hypertension, from baseline to 24 months
Change in Body Mass Index | Baseline; 12 months
  Change in body mass index between baseline and 12 months.
Change in Body Mass Index | Baseline; 24 months
  Change in body mass index between baseline and 24 months.
Change in waist circumference | Baseline; 12 months
  Change in waist circumference between baseline and 12 months
Change in waist circumference | Baseline; 24 months
  Change in waist circumference between baseline and 24 months
Change in fruit intake | Baseline; 12 months
  Change in reported number of servings of fruits consumed per week between baseline and 12 months
Change in fruit intake | Baseline; 24 months
  Change in reported number of servings of fruits consumed per week between baseline and 24 months
Change in vegetables intake | Baseline; 12 months
  Change in reported number of servings of vegetables consumed per week between baseline and 12 months
Change in vegetables intake | Baseline; 24 months
  Change in reported number of servings of vegetables consumed per week between baseline and 24 months
Change in minutes of physical exercise per week | Baseline; 12 months
  Change in minutes of physical exercise per week between baseline and 12 months
Change in minutes of physical exercise per week | Baseline; 24 months
  Change in minutes of physical exercise per week between baseline and 24 months
Reach of the intervention | 24 months
  Percentage of religious leaders attending educational seminar and mentorship groups of 240 invited and number of community members reporting having blood pressure measured in the past year
Effectiveness of the intervention | 24 months
  Percentage of community members initiating anti-hypertensive medications
Adoption of the intervention | 24 months
  Percentage of community members report being educated about blood pressure by religious leader in past 12 months
Maintenance of the intervention | 24 months
  Percentage of community members report hearing blood pressure discussed in religious context in past 12 months; self-efficacy for blood pressure
Mean change in community systolic blood pressure | Baseline; 24 months
  Before and 24 months after the intervention, investigators will estimate the true mean community BP by sampling 400 randomly selected adult community members (age ≥35 years) in each of the 20 communities.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Downs, MD, PhD, Principal Investigator — Weill Medical College of Cornell University; Robert N Peck, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Community, Wards, Mwanza, Geita, and Simiyu Regions, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
De-identified research data sets that document, support, and validate our research findings will be made available under appropriate data-sharing agreements after the main findings from the final research data set have been accepted for publication.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available at the time of manuscript publication.
Access Criteria: De-identified data on community blood pressures, including demographic and clinical data, will be made available under appropriate data-sharing agreements.